CLINICAL TRIAL: NCT00799552
Title: A Phase II, Multi-Center, Double-Masked, Randomized, Placebo Controlled, Study on the Safety and Efficacy of RX-10045 on the Signs and Symptoms of Dry Eye in Every Day Environmental Conditions and During Provocation Using the Controlled Adverse Environment (CAE) Model
Brief Title: Safety and Efficacy Study of RX-10045 on the Signs and Symptoms of Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resolvyx Pharmaceuticals, Inc (Industry)
Responsible Party: Per Gjorstrup, Chief Medical Officier, Resolvyx Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-004-03
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Dry Eye Syndrome
Keywords: Keratoconjunctivitis Sicca; Dry eye; Resolvin
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — isopropyl 5,12-hydroxypentadeca-8,10-dien-6,14-diynoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RX-10045 (Experimental)
  Interventions: Drug: RX-10045

INTERVENTIONS:
Drug: RX-10045 — RX-10045 eye drop
  Arms: RX-10045
Drug: Placebo — Placebo eye drop
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and efficacy of RX-10045 to placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Have provided written informed consent;
* Have a history of dry eye for at least 6 months prior to enrollment;
* Have a history of use or desire to use eye drops for dry eye symptoms within the past 6 months;
* Demonstrate a response when exposed to the CAE.

Exclusion Criteria:

* Have an on-going ocular infection, or active ocular inflammation
* Have worn contact lenses within 72 hours of Visit 1 or have anticipated use of contact lenses during the study;
* Have contact lens-induced dry eye;
* Have previously had laser in situ keratomileusis (LASIK) surgery;
* Be using or have anticipated use of temporary punctual plugs during the study;
* Have best corrected visual acuity > +0.7 in both eyes;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Have a known allergy and/or sensitivity to the test article or its components;
* Be currently using any medication known to cause ocular drying that is not used on a stable dosing regimen for at least 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining and integrated subject diary data | 28 days

SECONDARY OUTCOMES:
Changes in dry eye signs and symptoms | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Ophthalmic Research Associates, Andover, MA; John Lonsdale, MD, Principal Investigator — Central Maine Eye Care, Lewiston, ME; Joel Geffin, MD, Principal Investigator — The Eye Care Group, Waterbury, CT
Locations (1):
- ORA Clinical, Andover, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.resolvyx.com